CLINICAL TRIAL: NCT02916394
Title: Targeted Molecular Imaging of [68Ga]- Labelling Anti-IGF-1R Affibody Molecule in IGF-1R Overexpression Cancer Patients （Such as Colon Cancer、NSCLC and Gliomas）and Healthy Volunteers
Brief Title: In Vivo IGF-1R Molecular Imaging Using [68Ga]- Labelling Anti-IGF-1R Affibody Molecule
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yingying Sun, Chief, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14403
Record Dates: First submitted 2016-09-24; First posted 2016-09-27 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Molecular Imaging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 68Ga-NODAGA-ZIGF-1R:4：40：IGF-1R+++ (Experimental): Patients in this group had IGF-1R overexpression tumors and did not receive any treatment before this study.
  Interventions: Radiation: 68Ga-NODAGA-ZIGF-1R:4：40
- 68Ga-NODAGA-ZIGF-1R:4：40：IGF-1R++ (Experimental): Patients in this group had IGF-1R moderate expression tumors and did not receive any treatment before this study.
  Interventions: Radiation: 68Ga-NODAGA-ZIGF-1R:4：40
- 68Ga-NODAGA-ZIGF-1R:4：40：IGF-1R+ (Experimental): Patients in this group had IGF-1R low expression tumors and did not receive any treatment before this study.
  Interventions: Radiation: 68Ga-NODAGA-ZIGF-1R:4：40
- 68Ga-NODAGA-ZIGF-1R:4：40：healthy volunteers (Experimental): Patients in this group who are healthy volunteer.
  Interventions: Radiation: 68Ga-NODAGA-ZIGF-1R:4：40

INTERVENTIONS:
Radiation: 68Ga-NODAGA-ZIGF-1R:4：40 — No Intervention

SUMMARY:
The investigators developed [68Ga]-labelling Anti-IGF-1R Affibody Molecule as a targeted molecular imaging agent for noninvasive and repeatable detecting IGF-1R expression status.

DETAILED DESCRIPTION:
The goals of investigators are to evaluate the use of [68Ga]-labelling Anti-IGF-1R Affibody Molecule as a novel PET/CT radiotracer to monitor IGF-1R expression status. The investigators want to evaluate the use of [68Ga]-labelling Anti-IGF-1R Affibody Molecule in IGF-1R expression cancer imaging in adult cancer patients （colon cancer 、NSCLC、gliomas cancer patients）with different IGF-1R expression status.

ELIGIBILITY:
Inclusion Criteria:

1. Colon cancer, NSCLC and gliomas patients with pathological and gene detection results and did not receive any treatment
2. More than 18 years old
3. A life expectancy of at least 12 weeks
4. Presence of a malignant lesion within the chest of at least 0.5 cm diameter as measured by computed tomography (CT)
5. Written informed consent

Exclusion Criteria:

1. Could not get pathological and gene detection results
2. Pregnancy
3. do not want to write informed consent。

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
tumor SUV value of 68Ga-NODAGA-ZIGF-1R:4:40 PET/CT Imaging | after scanning(at time of imaging)
  To quantify the accumulation, a volume of interest using a 3D sphere, was placed over the tumor, lymph nodes and distant metastases avoiding necrosis, blood vessels and normal tissues as much as possible on a workstation (Advantage Workstation 4.6; GE Healthcare). The maximum standard uptake value (SUVmax) normalized to body weight (kBq/mL) was calculated within the region of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Baozhong Shen, Study Chair — The Fourth Hospital of Harbin Medical University
Locations (1):
- TOF-PET/CT/MR center of the Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided